CLINICAL TRIAL: NCT05698628
Title: Comparison Of Conservative Versus Early Distal Perfusion Strategy to Prevent Acute Limb Ischemia in Peripheral Venoarterial Extracorporeal Membrane Oxygenation Patients
Brief Title: Distal Perfusion Timing, Early or Conservative, to Prevent Limb Ischemia During Peripheral VA-ECMO
Acronym: DECIDE-ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Min-Seok Kim (Other)
Responsible Party: Sponsor-Investigator, Min-Seok Kim, Clinical Associate Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_2022_1691
Record Dates: First submitted 2023-01-12; First posted 2023-01-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: Extracorporeal Membrane Oxygenation; Limb ischemia; Cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preemptive distal perfusion group (Experimental): Distal perfusion catheterization will be done within 1 hour after VA-ECMO application.
  Interventions: Procedure: Distal perfusion catheterization
- Conventional distal perfusion group (Active Comparator): The conventional group will undergo distal perfusion catheterization at the time of limb ischemia sign.
  Interventions: Procedure: Distal perfusion catheterization

INTERVENTIONS:
Procedure: Distal perfusion catheterization — Distal perfusion catheterization will be done within 1 hour after the VA-ECMO application in the preemptive DPC group. The conventional DPC group will undergo distal perfusion catheterization at the time of limb ischemia sign.

SUMMARY:
Peripheral VA-ECMO is widely used in refractory cardiogenic shock patients as a salvage therapy. In most cases, the femoral artery and vein are used for the vascular approach. Large cannulas are usually used for proper oxygenation, which may cause peripheral limb ischemia. Distal perfusion catheterization (DPC) at the ipsilateral arterial cannula site is recommended to prevent distal limb ischemia. However, there is no consensus on the proper timing of DPC and additional invasive procedures may cause complications during VA-ECMO support. In this analysis, the investigators compare the clinical outcomes of distal limb ischemia complications between the conventional DPC group (DPC at the time of limb ischemia sign) and the preemptive DPC group (DPC at the time of VA-ECMO application).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 years old
* Refractory cardiogenic shock with peripheral VA-ECMO
* Informed consent

Exclusion Criteria:

* Unwilling or unable to obtain informed consent from the participant or substitute decision-maker
* Patients who are currently pregnant, postpartum period within 30 days or are breast-feeding
* VA-ECMO application for causes other than cardiogenic shock
* Severe coagulopathy
* Irreversible limb ischemia requiring interventional procedures or surgery at the time of VA-ECMO (previously diagnosed ASO(atherosclerosis obliterans) patients)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Limb ischemia | From date of randomization until the date of discharge or assessed up to 90 days
  Limb ischemia requiring surgical/percutaneous procedure or resulting necrosis or neurologic sequelae in the distal limb during hospitalization

SECONDARY OUTCOMES:
All-cause mortality | From date of randomization until the date of death from any cause, assessed up to 12 months
  All-cause of death
Successful ECMO weaning | From date of randomization until the date of discharge or assessed up to 90 days
  Having ECMO removed and not requiring further mechanical support because of recurring cardiogenic shock over the following 30 days
ECMO related complications | From date of randomization until the date of ECMO removal, assesed up to 90 days
  Bleeding, systemic thromboembolism, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Seok Kim, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No